CLINICAL TRIAL: NCT01837719
Title: A Randomized, 5-Period, Crossover Study in Healthy Subjects to Assess the Bioequivalence of Atazanavir When Co-Administered With Cobicistat as a Fixed Dose Combination Relative to the Single Agents Following a Light Meal, the Relative Bioavailability of Atazanavir When Co-Administered With Cobicistat as a Fixed Dose Combination Relative to the Single Agents Under Fasted Conditions, and the Effect of Food on the Bioavailability of Atazanavir in the Fixed Dose Combination
Brief Title: Bioequivalence Study of Individual Atazanavir and Cobicistat Compared With Atazanavir in Fixed-dose Combination With Cobicistat
Acronym: Atazanavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AI424-511
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Atazanavir Sulfate; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A: Atazanavir + Cobicistat coadministered (Experimental): Participants received a single dose of atazanavir, 300 mg as capsule, coadministered with cobicistat,150 mg as tablet, following a light meal on Day 1 or 8
  Interventions: Drug: Atazanavir; Drug: Cobicistat
- Treatment B: Atazanavir/Cobicistat FDC (Experimental): Participants received a single fixed-dose combination (FDC) of atazanavir, 300 mg/cobicistat, 150 mg, following a light meal on Day 1 or 8
  Interventions: Drug: Atazanavir/Cobicistat FDC
- Treatment C: Atazanavir + Cobicistat coadministered (Experimental): Participants received a single dose of atazanavir, 300 mg as capsule, coadministered with cobicistat,150 mg as tablet, in the fasted state on Day 15 or 22
  Interventions: Drug: Atazanavir; Drug: Cobicistat
- Treatment D: Atazanavir/Cobicistat FDC (Experimental): Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, in the fasted state on Day 15 or 22
  Interventions: Drug: Atazanavir/Cobicistat FDC
- Treatment E: Atazanavir/Cobicistat FDC (Experimental): Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, following a high-fat meal on Day 29
  Interventions: Drug: Atazanavir/Cobicistat FDC

INTERVENTIONS:
Drug: Atazanavir — 300-mg capsule
  Other Names: BMS-232632
  Arms: Treatment A: Atazanavir + Cobicistat coadministered; Treatment C: Atazanavir + Cobicistat coadministered
Drug: Cobicistat — 150-mg tablet
  Arms: Treatment A: Atazanavir + Cobicistat coadministered; Treatment C: Atazanavir + Cobicistat coadministered
Drug: Atazanavir/Cobicistat FDC — Atazanavir 300-mg/cobicistat 150-mg FDC tablet
  Arms: Treatment B: Atazanavir/Cobicistat FDC; Treatment D: Atazanavir/Cobicistat FDC; Treatment E: Atazanavir/Cobicistat FDC

SUMMARY:
The purpose of the study is to compare the pharmacokinetics and bioequivalence of atazanavir in a fixed-dose combination with cobicistat with that of atazanavir coadministered with cobicistat as single agents.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy men and women, ages 18 to 49 years
* Body mass index 18 to 32 kg/m^2, inclusive
* Women of childbearing potential (WOCBP) who were not pregnant or breastfeeding
* WOCBP and men who are sexually active with WOCBP must use acceptable contraceptive methods

Key Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) gastrointestinal tract disease
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal tract surgery (including cholecystectomy) that could have an impact on the absorption of study drug
* Donation of blood to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration (within 2 weeks for plasma only)
* Blood transfusion within 4 weeks of study drug administration
* Inability to tolerate oral medication, to be venipunctured, or to tolerate venous access
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination or electrocardiogram (ECG) findings, vital sign measurements, or results of clinical laboratory tests, beyond what is consistent with the target population
* Any of the following 12-lead ECG findings prior to study drug administration, confirmed by repeat testing

  * PR ≥210 msec
  * QRS ≥120 msec
  * QT ≥500 msec
  * QTcF ≥450 msec
* 2nd- or 3rd-degree A-V block or clinically relevant abnormalities in ECG findings
* Positive result on urine screening for drugs of abuse
* Positive result on blood screening for hepatitis C antibody, hepatitis B surface antigen, or HIV-1 or -2 antibody
* Laboratory test results indicating levels outside of the ranges specified below:

  * Alanine aminotransferase >upper limit of normal (ULN)
  * Aspartate aminotransferase >ULN
  * Total bilirubin >ULN
  * Serum creatinine >ULN

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Inc., Austin, Texas, United States

REFERENCES:
- [Derived] Sevinsky H, Tao X, Wang R, Ravindran P, Sims K, Xu X, Jariwala N, Bertz R. A randomized trial in healthy subjects to assess the bioequivalence of an atazanavir/cobicistat fixed-dose combination tablet versus administration as separate agents. Antivir Ther. 2015;20(5):493-500. doi: 10.3851/IMP2913. Epub 2014 Oct 31. PMID 25361436

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 149 patients were enrolled and 64 randomized to 1 of 8 treatment sequences (ABCDE, ABDCE, BACDE, BADCE, ABCD, ABDC, BACD, or BADC), with a 7-day washout period between treatments. Approximately 32 were to be discharged after Period 4, based on treatment sequence. Those remaining were to continue to and be discharged at end of Period 5.
Groups:
- All Participants Who Received Treatment: All participants who received atazanavir with cobicistat in 1 of 8 treatment sequences (ABCDE, ABDCE, BACDE, BADCE, ABCD, ABDC, BACD, or BADC). Treatment A: Participants received a single dose of atazanavir, 300 mg as capsule, coadministered with cobicistat, 150 mg as tablet, following a light meal on Day 1 or 8. Treatment B: Participants received a single fixed-dose combination (FDC) of atazanavir, 300 mg/cobicistat, 150 mg, following a light meal on Day 1 or 8. Treatment C: Participants received a single dose of atazanavir, 300 mg as capsule, coadministered with cobicistat,150 mg as tablet, in the fasted state on Day15 or 22. Treatment D: Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, in the fasted state on Day 15 or 22. Treatment E: Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, following a high-fat meal on Day 29.
Period: Period 1: Days 1-7 (Treatment A or B)
Arm/Group | All Participants Who Received Treatment
Started | 64 (Received treatment)
Completed | 64
Not Completed | 0
Period: Period 2: Days 8-14 (Treatment B or A)
Arm/Group | All Participants Who Received Treatment
Started | 64
Completed | 63
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period 3: Days 15-21 (Treatment C or D)
Arm/Group | All Participants Who Received Treatment
Started | 63
Completed | 63
Not Completed | 0
Period: Period 4: Days 22-28 (Treatment D or C)
Arm/Group | All Participants Who Received Treatment
Started | 63
Completed | 63 (Number finishing period; 32 patients were discharged following Period 4, as per protocol)
Not Completed | 0
Period: Period 5: Days 29-31 (Treatment E)
Arm/Group | All Participants Who Received Treatment
Started | 31 (Reflects the 31 patients remaining after 32 were discharged at the end of Period 4, as per protocol)
Completed | 30
Not Completed | 1
Not completed — Poor compliance/noncompliance | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- All Participants Who Received Treatment: All participants who received atazanavir with cobicistat in 1 of 8 treatment sequences (ABCDE, ABDCE, BACDE, BADCE, ABCD, ABDC, BACD, or BADC). Treatment A: Participants received a single dose of atazanavir, 300 mg as capsule, coadministered with cobicistat,150 mg as tablet, following a light meal on Day 1 or 8. Treatment B: Participants received a single fixed-dose combination (FDC) of atazanavir, 300 mg/cobicistat, 150 mg, following a light meal on Day 1 or 8. Treatment C: Participants received a single dose of atazanavir, 300 mg as capsule, coadministered with cobicistat,150 mg as tablet, in the fasted state on Day 15 or 22. Treatment D: Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, in the fasted state on Day15 or 29. Treatment E: Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, following a high-fat meal on Day 29.
Arm/Group | All Participants Who Received Treatment
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 29
  Black | 33
  Asian | 2
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Atazanavir
Description: Blood samples for plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. Cmax was derived from plasma concentration versus time data.
Time Frame: Days 1, 8, 15, 22, and 29 (predose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 12, and 16 hours postdose); Days 2, 9, 16, 23, and 30 (24, 30, and 36 hours postdose); Days 3, 10, 17, 24, and 31 (48 hours postdose)
Population: All participants who received any study medication and had any available concentration-time data. All available derived pharmacokinetic (PK) parameter values were included in the PK data set and reported, but only those with adequate PK profiles were included in the summary statistics and statistical analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
ng/mL | 3832 (39) | 4104 (32) | 2585 (45) | 2941 (44) | 2545 (43)
Statistical Analysis 1: Comparison: Treatment A: Atazanavir + Cobicistat Coadministered vs Treatment B: Atazanavir/Cobicistat FDC; To demonstrate bioequivalence for atazanavir between the test (Treatment B) and reference (Treatment A) formulations, a linear mixed-effects model was applied to the natural logarithms of atazanavir Cmax, with treatment, period, and sequence as fixed effects, and participant (sequence) as a random effect; Test type: Non-Inferiority or Equivalence — Bioequivalence was concluded if the 90% CI for the ratios of geometric means of the test formulation (fixed-dose combination [FDC] tablet of 300/150 mg atazanavir/cobicistat) to the reference formulation (300-mg atazanavir capsule coadministered with 150-mg cobicistat) were contained within 0.80 to 1.25 for atazanavir Cmax, area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC[0-T]) and AUC from time 0 to infinity. (AUC[0-T]); Mixed Models Analysis; Geometric mean ratio = 1.073, 90% CI 2-sided [1.012 to 1.137] — Geometric mean ratio is calculated as Treatment B/Treatment A
Statistical Analysis 2: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment D: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of a light meal and the fasted state on the natural logarithms of exposure of atazanavir when given as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.423, 90% CI 2-sided [1.273 to 1.590] — Geometric mean ratio was calculated as Treatment B/Treatment D
Statistical Analysis 3: Comparison: Treatment C: Atazanavir + Cobicistat Coadministered vs Treatment D: Atazanavir/Cobicistat FDC; To assess the relative bioavailability of atazanavir under fasted (Treatment D) versus fed (Treatment C) states, a linear mixed-effects model was applied to the natural logarithms of atazanavir Cmax with treatment, period, and sequence as fixed effects and participant (sequence) as a random effect; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.137, 90% CI 2-sided [1.000 to 1.292] — Geometric mean ratio is calculated as Treatment D/Treatment C
Statistical Analysis 4: Comparison: Treatment D: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of a high fat meal and the fasted state on the natural logarithms of exposure of atazanavir when given as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.862, 90% CI 2-sided [0.701 to 1.059] — Geometric mean ratio is calculated as Treatment E/Treatment D
Statistical Analysis 5: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of high fat and light meals on the natural logarithms of exposure of atazanavir when given as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.643, 90% CI 2-sided [0.545 to 0.759] — Geometric mean ratio is calculated as Treatment E/Treatment B

2. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Time of Last Quantifiable Concentration (AUC[0-T]) and From Time 0 to Infinity (AUC[INF]) for Atazanavir
Description: Blood samples for plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. AUC(0-T) and AUC(INF) were derived from plasma concentration versus time data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
ng*h/mL
  AUC(0-T) | 32775 (38) | 34905 (32) | 25017 (46) | 27875 (41) | 25873 (40)
  AUC(0-INF) | 33523 (39) | 35673 (32) | 25547 (47) | 28378 (42) | 26510 (40)
Statistical Analysis 1: Comparison: Treatment A: Atazanavir + Cobicistat Coadministered vs Treatment B: Atazanavir/Cobicistat FDC; Bioequivalence was concluded if the 90% confidence intervals for the ratios of geometric means of the test formulation (FDC tablet of 300/150 mg atazanavir/cobicistat) to the reference formulation (300-mg atazanavir capsule coadministered with 150-mg cobicistat) were contained within 0.80 to 1.25 for atazanavir Cmax, AUC(0-T) and AUC(INF); Test type: Non-Inferiority or Equivalence — To demonstrate bioequivalence for atazanavir between the test (Treatment B) and reference (Treatment A) formulations, a linear mixed-effects model was applied to the natural logarithms of atazanavir AUC(0-T), with treatment, period, and sequence as fixed effects, and participant (sequence) as a random effect; Mixed Models Analysis; Geometric mean ratio = 1.065, 90% CI 2-sided [1.012 to 1.120] — Geometric mean ratio for AUC(0-T) is calculated as Treatment B/Treatment A
Statistical Analysis 2: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment D: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and patient as a random effect was used to estimate the effect of a light meal and the fasted state on the natural logarithms of exposure of atazanavir when administered as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.275, 90% CI 2-sided [1.166 to 1.393] — Geometric mean ratio for AUC(0-T) was calculated as Treatment B/Treatment D
Statistical Analysis 3: Comparison: Treatment C: Atazanavir + Cobicistat Coadministered vs Treatment D: Atazanavir/Cobicistat FDC; To assess the relative bioavailability of atazanavir under fasted (Treatment D) versus fed (Treatment C) states, a linear mixed-effects model was applied to the natural logarithms of atazanavir AUC(0-T) with treatment, period, and sequence as fixed effects and participant (sequence) as a random effect; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.113, 90% CI 2-sided [0.993 to 1.248] — Geometric mean ratio for AUC(0-T) is calculated as Treatment D/Treatment C
Statistical Analysis 4: Comparison: Treatment D: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and participant as a random effect will be used to estimate the effect of a high fat meal and the fasted state on the natural logarithms of exposure of atazanavir when given as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.950, 90% CI 2-sided [0.804 to 1.122] — Geometric mean ratio of AUC(0-T) was calculated as Treatment E/Treatment D
Statistical Analysis 5: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and participant as a random effect will be used to estimate the effect of high fat and light meals on the natural logarithms of exposure of atazanavir when given as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.746, 90% CI 2-sided [0.655 to 0.849] — Geometric mean ratio of AUC(0-T) was calculated as Treatment E/Treatment B
Statistical Analysis 6: Comparison: Treatment A: Atazanavir + Cobicistat Coadministered vs Treatment B: Atazanavir/Cobicistat FDC; To demonstrate bioequivalence for atazanavir between the test (Treatment B) and reference (Treatment A) formulations, a linear mixed-effects model was applied to the natural logarithms of atazanavir AUC(0-INF), with treatment period and sequence as fixed effects, and patient (sequence) as a random effect; Test type: Non-Inferiority or Equivalence — Bioequivalence was concluded if the 90% confidence intervals for the ratios of geometric means of the test formulation (FDC tablet of 300/150 mg atazanavir/cobicistat) to the reference formulation (300-mg atazanavir capsule coadministered with 150-mg cobicistat) were contained within 0.80 to 1.25 for atazanavir Cmax, AUC(0-T) and AUC(INF); Mixed Models Analysis; Geometric mean ratio = 1.064, 90% CI [1.011 to 1.120] — Geometric mean ration for AUC(INF) is calculated as Treatment B/Treatment A
Statistical Analysis 7: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment D: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and participant as a random effect was used to estimate the effect of a light meal and fthe fasted state on the natural logarithms of exposure of atazanavir when given as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.280, 90% CI 2-sided [1.171 to 1.398] — Geometric mean ratio for AUC(INF) was calculated as Treatment B/Treatment D
Statistical Analysis 8: Comparison: Treatment C: Atazanavir + Cobicistat Coadministered vs Treatment D: Atazanavir/Cobicistat FDC; To assess the relative bioavailability of atazanavir under fasted (Treatment D) versus fed (Treatment C) states, a linear mixed-effects model was applied to the natural logarithms of atazanavir AUC(0-INF) with treatment, period, and sequence as fixed effects and participant (sequence) as a random effect; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.110, 90% CI 2-sided [0.991 to 1.244] — Geometric mean ratio of AUC(INF) was calculated as Treatment D/Treatment C
Statistical Analysis 9: Comparison: Treatment D: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.956, 90% CI 2-sided [0.810 to 1.128] — Geometric mean of AUC(INF) was calculated as Treatment E/Treatment D
Statistical Analysis 10: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and participant as a random effect was used to estimate the effect of high fat and light meals on the natural logarithms of exposure of atazanavir when administered as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.749, 90% CI 2-sided [0.658 to 0.852] — Geometric mean ratio of AUC(INF) was calculated as Treatment E/Treatment B

3. Secondary Outcome: Number of Participants Who Died and With Serious Adverse Events (SAEs)
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant who receives an investigational product and that does not necessarily have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product. An SAE is any untoward medical occurrence that at any dose results in death; is life-threatening; or requires or prolongs inpatient hospitalization.
Time Frame: On Day 24 or 31
Population: All participants who received at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 64 | 64 | 64 | 63 | 30
Participants
  Deaths | 0 | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Marked Abnormalities in Results of Clinical Laboratory Tests
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRx=pretreatment; h=high; hpf=high power field. Abnormal criteria: Leukocytes, low (*10^3 c/uL): <0.85*preRx if preRx<LLN; <0.9*LLN if LLN≤preRx≤ULN;< 0.9*LLN if preRx=missing;<LLN if preRX>ULN. Neutrophils, low (*10^3 c/uL): <0.85*preRx if preRx<1.5; <1.5 if preRx=missing; <1.5 if preRx ≥1.5. Bilirubin, h (mg/dL): >1.1* ULN if preRx≤ULN; >1.1*ULN if preRx=missing; >1.25*preRx if preRx>ULN. Bilirubin, h (mg/dL): >1.1* ULN if preRx≤ULN; >1.1*ULN if preRx=missing; >1.25*preRx if preRx>ULN. Blood, urine, h: ≥2*preRx if preRx≥1; ≥2 if preRx <1; ≥2 if preRx=missing. RBCs/WBCs, h (hpf): ≥2 if preRx=missing ≥2 if preRx<2 ≥4 if preRx ≥2. Creatine kinase, h (U/L): >1.5*preRx if preRx>ULN; >1.5*ULN if preRx≤ULN; >1.5*ULN if preRx=missing; AST, h (U/L): >1.25* preRx if preRx>ULN; >1.25*ULN if preRx≤ULN; >1.25*ULN if preRx=missing. Lactate dehydrogenase, h (U/L): >1.25*ULN if preRx≤ULN; >1.25*ULN if preRx=missing; >1.5*preRx if preRx>ULN.
Time Frame: At Screening and on Days -1,4, 11, 18, and 31 (study discharge)
Population: All participants who received at least 1 dose of study drug and had laboratory test results available.
Measure: Number; unit: Participants
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 63 | 63 | 63 | 30
Participants
  Leukocytes (low) | 3 | 2 | 3 | 1 | 1
  Neutrophils, absolute (low) | 2 | 4 | 3 | 2 | 1
  Bilirubin, total (high) | 1 | 0 | 0 | 3 | 4
  Bilirubin, direct | 0 | 0 | 0 | 1 | 1
  Blood, urine (high) | 1 | 0 | 0 | 1 | 1
  Red blood cells (RBC), urine (high) | 1 | 0 | 0 | 0 | 1
  White blood cells (WBC), urine (high) | 2 | 0 | 0 | 3 | 2
  Creatine kinase (high) | 0 | 1 | 1 | 0 | 0
  Aspartate aminotransferase (AST) (high) | 0 | 0 | 1 | 0 | 0
  Lactate dehydrogenase (high) | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With Out-of-range Intervals on Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded at predose and 4 hours post dose at screening, Days -1, 1, 8 15, 22, 29 and study discharge. ECGs were recorded after the patient had been supine for at least 5 minutes. All ECG readings post dosing (including unscheduled) were included.
Time Frame: At screening; on Day -1; predose and 4 hours postdose on Days 1, 18, 15, 22, and 29; and at study discharge (Day 31)
Population: All participants who received at least 1 dose of study medication and were evaluable.
Measure: Number; unit: Participants
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 63 | 63 | 63 | 30
Participants
  PR interval >210 msec | 0 | 0 | 0 | 1 | 0
  QRS interval >120 msec | 1 | 1 | 0 | 0 | 0
  QT interval >500 msec | 0 | 0 | 0 | 0 | 0
  QTcF>450 msec | 1 | 0 | 0 | 0 | 0

6. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Atazanavir
Description: Blood samples for plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. Tmax was derived from plasma concentration versus time data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Groups:
- Treatment D: Atazanavir/Cobicistat FDC: Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, in the fasted state on Day15 or 22
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
Hours | 3.00 (39) [2.0 to 5.5] | 2.50 [2.0 to 4.05] | 2.00 [1.00 to 8.00] | 2.00 [1.00 to 6.00] | 3.54 [2.00 to 8.02]

7. Secondary Outcome: Observed Concentration at 24 Hours (C24) of Atazanavir
Description: Blood samples for plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. C24 was derived from plasma concentration versus time data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
ng/mL | 416 (58) | 449 (52) | 295 (63) | 337 (56) | 398 (45)
Statistical Analysis 1: Comparison: Treatment A: Atazanavir + Cobicistat Coadministered vs Treatment B: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and patient as random effect will be used to estimate the effect of a light meal and the fasted state on the natural logarithms of exposure of atazanavir when administered as a fixed-dose combination; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.084, 90% CI 2-sided [1.014 to 1.158] — Geometric mean ratio was calculated as Treatment B/Treatment A
Statistical Analysis 2: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment D: Atazanavir/Cobicistat FDC; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.349, 90% CI 2-sided [1.215 to 1.498] — Geometric mean ratio of C24 was calculated as Treatment B/Treatment D
Statistical Analysis 3: Comparison: Treatment C: Atazanavir + Cobicistat Coadministered vs Treatment D: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and patient as random effect will be used to estimate the effect of a light meal and the fasted state on the natural logarithms of exposure of atazanavir when administered as an FDC; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.144, 90% CI [1.006 to 1.300] — Geometric mean ratio was calculated as Treatment D/Treatment C
Statistical Analysis 4: Comparison: Treatment D: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 1.231, 90% CI 2-sided [1.023 to 1.483] — Geometric mean ratio was calculated as Treatment E/Treatment D
Statistical Analysis 5: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.912, 90% CI [0.789 to 1.054] — Geometric mean ratio was calculated as Treatment E/Treatment B

8. Secondary Outcome: Apparent Terminal Half-life (T-HALF) of Atazanavir
Description: Blood samples for testing plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. T-HALF was derived from plasma concentration versus time data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
Hours | 7.54 (2.91) | 7.50 (2.60) | 7.25 (2.49) | 7.21 (2.28) | 7.14 (2.99)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Cobicistat
Description: Blood samples for testing plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. Cmax was derived from plasma concentration versus time data.
Time Frame: Days 1, 8, 15, 22, and 29 (1,2, 2.5, 3, 4, 5, 6, 8, 12, and 16 hours postdose); Days 2, 9, 16, 23, and 30 (24 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment D: Atazanavir/Cobicistat FDC: Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, in the fasted state on Day15 or22
- Treatment E: Atazanavir/Cobicistat FDC: Participants received a single FDC dose of atazanavir, 300 mg/cobicistat, 150 mg, following a high fat meal on Day 29
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
ng/mL | 1321 (32) | 1348 (29) | 952 (39) | 1033 (38) | 1060 (32)
Statistical Analysis 1: Comparison: Treatment A: Atazanavir + Cobicistat Coadministered vs Treatment B: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and patient as random effect will be used to estimate the effect of a light meal and the fasted state on the natural logarithms of exposure of cobicistat when administered as a fixed-dose combination; Test type: Superiority or Other; Geometric mean ratio = 1.023, 90% CI 2-sided [0.991 to 1.057] — Geometric mean ratio was calculated as Treatment B/Treatment A
Statistical Analysis 2: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment D: Atazanavir/Cobicistat FDC; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 1.305, 90% CI 2-sided [1.215 to 1.402] — Geometric mean ratio was calculated as Treatment B/Treatment D
Statistical Analysis 3: Comparison: Treatment C: Atazanavir + Cobicistat Coadministered vs Treatment D: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effect and patient as random effect will be used to estimate the effect of a light meal and the fasted state on the natural logarithms of exposure of atazanavir cobicistat; Test type: Superiority or Other; Geometric mean ratio = 1.085, 90% CI 2-sided [0.925 to 1.273] — Geometric mean ratio was calculated as Treatment D/Treatment C
Statistical Analysis 4: Comparison: Treatment D: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 1.040, 90% CI 2-sided [0.937 to 1.154] — Geometric mean ratio was calculated asTreatment E/Treatment D
Statistical Analysis 5: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Geometric mean ratio = 0.784, 90% CI 2-sided [0.717 to 0.858] — Geometric mean ratio was calculated as Treatment E/Treatment B

10. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Cobicistat
Description: Blood samples for testing plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. Tmax was derived from plasma concentration versus time data.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
Hours | 2.52 [1.00 to 5.00] | 2.52 [1.00 to 5.00] | 2.00 [1.00 to 5.00] | 2.00 [1.00 to 5.00] | 4.00 [1.00 to 12.00]

11. Secondary Outcome: Area Under the Concentration Curve From Time 0 to Time of Last Quantifiable Concentration (AUC[0-T]) and Area Under the Concentration Curve From Time 0 to Infinity (AUC[INF]) of Cobicistat
Description: Blood samples for testing plasma concentrations were obtained at predose and at specific timepoints up to 48 hours after dosing on Days 1, 8, 15, 22, and 29. AUC(0-T) and AUC(INF) were derived from plasma concentration versus time data.
Time Frame: as for outcome 9
Population: All participants who received any study medication and had any available concentration-time data. All available derived pharmacokinetic (PK) parameter values were included in the PK data set and reported, but only those with adequate PK profiles were included in the summary statistics and statistical analysis. n=evaluable participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 30
ng*h/mL
  AUC(0-T) | 8738 (42) | 8866 (38) | 6541 (47) | 7204 (44) | 7916 (39)
  AUC(INF) (n=63, 62, 63, 63, 28) | 9045 (45) | 9178 (41) | 7884 (45) | 7408 (46) | 8298 (39)
Statistical Analysis 1: Comparison: Treatment A: Atazanavir + Cobicistat Coadministered vs Treatment B: Atazanavir/Cobicistat FDC; A linear mixed-effect model was applied to the natural logarithms of cobicistat AUC(0-T) with treatment, period, and sequence as fixed effects and participant (sequence) as a random effect; Test type: Superiority or Other; Geometric mean ratio = 1.019, 90% CI 2-sided [0.983 to 1.057] — Geometric mean ratio of AUC(0-T) was calculated as Treatment B/Treatment A
Statistical Analysis 2: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment D: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of a light meal and the fasted state on the natural logarithms of exposure of cobicistat when given as an FDC; Test type: Superiority or Other; Geometric mean ratio = 1.232, 90% CI [1.141 to 1.331] — Geometric mean ratio of AUC(0-T) was calculated as Treatment B/Treatment D
Statistical Analysis 3: Comparison: Treatment C: Atazanavir + Cobicistat Coadministered vs Treatment D: Atazanavir/Cobicistat FDC; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 1.102, 90% CI 2-sided [0.929 to 1.307] — Geometric mean ratio of AUC(0-T) was calculated as Treatment D/Treatment C
Statistical Analysis 4: Comparison: Treatment D: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of a high fat meal and the fasted state on the natural logarithms of exposure of cobicistat when given as an FDC; Test type: Superiority or Other; Geometric mean ratio = 1.127, 90% CI [1.017 to 1.248] — Geometric mean ratio of AUC(0-T) was calculated asTreatment E/Treatment D
Statistical Analysis 5: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of a high fat meal and a light meal on the natural logarithms of exposure of cobicistat when given as an FDC; Test type: Superiority or Other; Geometric mean ratio = 0.890, 90% CI 2-sided [0.825 to 0.960] — Geometric mean ratio of AUC(0-T) was calculated asTreatment E/Treatment B
Statistical Analysis 6: Comparison: Treatment A: Atazanavir + Cobicistat Coadministered vs Treatment B: Atazanavir/Cobicistat FDC; To demonstrate bioequivalence for atazanavir between the test (Treatment B) and reference (Treatment A) formulations, a linear mixed-effects model was applied to the natural logarithms of atazanavir AUC(0-INF), with treatment, period, and sequence as fixed effects, and participant (sequence) as a random effect; Test type: Non-Inferiority or Equivalence — Bioequivalence was concluded if the 90% CI for the ratios of geometric means of the test formulation (FDC tablet of 300/150 mg atazanavir/cobicistat) to the reference formulation (300-mg atazanavir capsule coadministered with 150-mg cobicistat) were contained within 0.80 to 1.25 for atazanavir Cmax, AUC(0-T), and AUC(INF); Geometric mean ratio = 1.019, 90% CI 2-sided [0.982 to 1.058] — Geometric mean ratio of AUC(INF) was calculated as Treatment B/Treatment A
Statistical Analysis 7: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment D: Atazanavir/Cobicistat FDC; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; Geometric mean ratio = 1.240, 90% CI 2-sided [1.148 to 1.340] — Geometric mean ratio of AUC(INF) was calculated as Treatment B/Treatment D
Statistical Analysis 8: Comparison: Treatment C: Atazanavir + Cobicistat Coadministered vs Treatment D: Atazanavir/Cobicistat FDC; A linear mixed-effect model was applied to the natural logarithms of cobicistat AUC(INF) with treatment, period, and sequence as fixed effects and participant (sequence) as a random effect; Test type: Superiority or Other; Geometric mean ratio = 0.976, 90% CI 2-sided [0.886 to 1.075] — Geometric mean ratio of AUC(INF) was calculated as Treatment D/Treatment C
Statistical Analysis 9: Comparison: Treatment D: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of a high fat meal and fasted on the natural logarithms of exposure of cobicistat when given as an FDC; Test type: Superiority or Other; Geometric mean ratio = 1.116, 90% CI 2-sided [1.012 to 1.231] — Geometric mean ratio of AUC(INF) was calculated as Treatment E/Treatment D
Statistical Analysis 10: Comparison: Treatment B: Atazanavir/Cobicistat FDC vs Treatment E: Atazanavir/Cobicistat FDC; A linear mixed-effect model with treatment as fixed effects and participant as a random effect will be used to estimate the effect of a high fat meal and light meal on the natural logarithms of exposure of atazanavir when given as an FDC; Test type: Superiority or Other; Geometric mean ratio = 0.904, 90% CI 2-sided [0.836 to 0.978] — Geometric mean ratio of AUC(INF) was calculated as Treatment E/Treatment B

12. Secondary Outcome: T-HALF of Cobicistat
Description: as for outcome 8
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Number analyzed (Participants) | 63 | 62 | 61 | 63 | 28
Hours | 4.34 (1.45) | 4.33 (1.42) | 4.23 (1.32) | 4.09 (1.20) | 4.27 (1.39)

ADVERSE EVENTS:
Groups:
- Treatment A: Atazanavir + Cobicistat Coadministered: Participants received a single dose of atazanavir, 300 mg as capsule, coadministered with cobicistat, 150 mg as tablet, following a light meal on Day 1 or 8.
Arm/Group | Treatment A: Atazanavir + Cobicistat Coadministered | Treatment B: Atazanavir/Cobicistat FDC | Treatment C: Atazanavir + Cobicistat Coadministered | Treatment D: Atazanavir/Cobicistat FDC | Treatment E: Atazanavir/Cobicistat FDC
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 0/63 | 0/63 | 0/31
Other Adverse Events (participants affected / at risk) | 1/64 | 3/64 | 0/63 | 0/63 | 0/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment A: Atazanavir + Cobicistat Coadministered (N=64) | Treatment B: Atazanavir/Cobicistat FDC (N=64) | Treatment C: Atazanavir + Cobicistat Coadministered (N=63) | Treatment D: Atazanavir/Cobicistat FDC (N=63) | Treatment E: Atazanavir/Cobicistat FDC (N=31)
Dizziness (Nervous system disorders) | 1/63 | 3/63 | 0 | 0 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.